CLINICAL TRIAL: NCT03185793
Title: Dose-finding and Safety Study of SHR4640 in Subjects With Hyperuricemia (Asymptomatic and Gout)
Brief Title: Dose-finding and Safety Study of SHR4640 in Subjects With Hyperuricemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR4640-201
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Hyperuricemia
Keywords: SHR4640, Phase II, monotherapy, dose-finding
MeSH Terms: conditions — Hyperuricemia | interventions — ruzinurad; Benzbromarone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): placebo for 5 weeks
  Interventions: Drug: Placebo
- 2.5mg SHR4640 (Experimental): SHR4640 for 5 weeks
  Interventions: Drug: SHR4640
- 5mg SHR4640 (Experimental): SHR4640 for 5 weeks
  Interventions: Drug: SHR4640
- 10mg SHR4640 (Experimental): SHR4640 for 5 weeks
  Interventions: Drug: SHR4640
- 50mg benzbromarone (Active Comparator): Benzbromarone for 5 weeks
  Interventions: Drug: benzbromarone

INTERVENTIONS:
Drug: Placebo — Placebo once daily for 5 weeks
  Arms: Placebo
Drug: SHR4640 — 1mg SHR4640 once daily for a week, 2.5mg, 5mg or 10mg SHR4640 once daily for 4 weeks
  Arms: 10mg SHR4640; 2.5mg SHR4640; 5mg SHR4640
Drug: benzbromarone — 25mg benzbromarone once daily for a week, 50mg benzbromarone once daily for 4 weeks
  Arms: 50mg benzbromarone

SUMMARY:
The objective of the study is to assess efficacy and safety of SHR4640 in subjects with hyperuricemia.

ELIGIBILITY:
Inclusion Criteria:

1. 18-70 years, male or female;
2. Subject meets one of the following conditions:

1) Subject with a history of gout has a serum uric acid ≥480μmol/l at screening; 2) Subject with a history of hyperuricemia has a serum uric acid ≥540μmol/l at screening, and requiring long-term uric acid-lowering therapy per the investigator's judgment; 3) Subject with a history of hyperuricemia has a serum uric acid≥480μmol/l at screening, on stable treatment for hypertensive, hyperlipidemia or diabetes for at least 3 month, and requiring long-term uric acid-lowering therapy per the investigator's judgment; 3. 18kg/m2≤ BMI ≤32kg/m2.

Exclusion Criteria:

1. Subject who is pregnant or breastfeeding;
2. Alanine aminotransferase or Aspartate aminotransferase or total bilirubin>1.5 upper normal limit;
3. Estimated glomerular filtration rate (MDRD formula) ˂60ml/min;
4. HbA1c˃8%;
5. Subject with known hypersensitivity or allergy to SHR4640 or any component of SHR4640;
6. Subject with a history of malignancy;
7. Subject with a history of urolithiasis, or positive findings on ultrasound examination at screen
8. Subject within the last 3months has: myocardial infarction, angina, percutaneous transluminal coronary angioplasty, coronary artery bypass grafting, cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage, or transient ischemia attack;
9. Subject has acute gout flares within 2 weeks before randomization;
10. Subject who is taking any other urate-lowering medication (allopurinol, febuxostat, probenecid and benzbromarone) that is indicated within 2 weeks before randomization and can not stop during the study;
11. Subject who is taking more than 100mg once daily or unstable dosage aspirin within 2 weeks before randomization and can not stop during the study;
12. Subject who is taking any diuretic within 2 weeks before randomization and can not stop during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2017-07-20 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a serum uric level≤360μmol/l. | Week 5

SECONDARY OUTCOMES:
Actual change from baseline in serum uric level. | Week 5
Percentage change from baseline in serum uric level . | Week 5
Rate of gout flares requiring treatment. | Up to week 5
Incidence of gout flares requiring treatment. | Up to week 5
Proportion of subjects with a serum uric level≤360μmol/l | At week1, 2, 3 and 4
Proportion of subjects with a serum uric level consistent ≤360μmol/l | At week 3, 4 and 5
Actual change from baseline in serum uric level | At week 1, 2, 3 and 4
Percentage change from baseline in serum uric level | At week 1, 2, 3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, Principal Investigator — RenJi Hospital
Locations (1):
- Jiangsu Hengrui Medicine Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin Y, Chen X, Ding H, Ye P, Gu J, Wang X, Jiang Z, Li D, Wang Z, Long W, Li Z, Jiang G, Li X, Bi L, Jiang L, Wu J, Guo L, Cai X, Lu X, Chen Q, Chen H, Peng A, Zuo X, Ning R, Zhang Z, Tai Y, Zhang T, Bao C. Efficacy and safety of a selective URAT1 inhibitor SHR4640 in Chinese subjects with hyperuricaemia: a randomized controlled phase II study. Rheumatology (Oxford). 2021 Nov 3;60(11):5089-5097. doi: 10.1093/rheumatology/keab198. PMID 33693494